CLINICAL TRIAL: NCT05912777
Title: Comparison of a 3D Reconstruction of the Knee Based on MRI With a 3D Reconstruction of the Knee Based on Scanner - Exploratory Study
Brief Title: 3D Reconstruction of the Knee Based on MRI
Acronym: IMAGENOU3D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00531-44
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scanner Arm (Experimental): A scanner must be performed by Patients
  Interventions: Radiation: Scanner

INTERVENTIONS:
Radiation: Scanner — Scanner to be performed by patients

SUMMARY:
ACL tear is a pathology of the knee quite common in athletes mainly caused by a twisting movement. The diagnosis of ACL tear can be confirmed by MRI (magnetic resonance imaging). This method makes it possible to visualize the inside of the knee and to diagnose lesions associated with rupture of the ACL (in particular meniscal lesions).

Obtaining a 3D model of patients' joints from a imaging is of growing interest to plan the gesture in preoperative but also to evaluate this gesture postoperatively. In orthopedic surgery, the baseline preoperative imaging is MRI. However, 3D models are generally obtained from a scanner-like imaging.

In this context, obtaining a 3D model from MRI imaging would make it possible to have a model that fits into the care pathway patients, without subjecting them to irradiation and visualizing anatomical structures not visible on CT.

However, the geometric precision and the reproducibility of the 3D reconstructions of joints reconstructed from an MRI remains unknown and must be evaluated to consider their clinical use.

DETAILED DESCRIPTION:
Rupture of the anterior cruciate ligament (ACL) is a pathology of the knee quite common in athletes. The main cause of an ACL tear is, in the majority of cases, an indirect trauma, caused by a twisting movement (example: the foot remains blocked on the ground while the knee rotates in or out).

Sometimes the clinical examination of the ACL tear may not be conclusive.This is usually the case when the patient's knee swelling is too large and that clinical tests are then difficult to carry out. The diagnosis of ACL tear can therefore be confirmed by MRI (magnetic resonance imaging). This method makes it possible to visualize the inside of the knee. In addition, the realization of the MRI will also help to diagnose lesions associated with rupture of the ACL and in particular meniscal lesions. This exam has become indispensable and is carried out in the vast majority of cases.

Obtaining a 3D model of patients' joints from a imaging is of growing interest. These 3D models allow particular to plan the gesture in preoperative but also to evaluate this gesture postoperatively. In orthopedic surgery, for patients suffering from an ACL tear, the baseline preoperative imaging is MRI. However, 3D models are generally obtained from a scanner-like imaging. This imagery has the advantage of presenting a very good definition of bone tissue but it is not part, for a large number of patients, routine preoperative imaging. It is irradiating and does not allow easy highlighting of other structures such as cartilage or menisci.

In this context, obtaining a 3D model from MRI imaging would make it possible to have a model that fits into the care pathway patients, without subjecting them to irradiation and visualizing anatomical structures not visible on CT.

However, the geometric precision and the reproducibility of the 3D reconstructions of joints reconstructed from an MRI remains unknown and must be evaluated to consider their clinical use. This is the purpose of this research.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged between ≥ 18 and ≤ 45 years old
* Patient eligible for ACL reconstruction
* Patient with an MRI performed at the SANTY orthopedic center or according to the protocol defined by the radiologists of the orthopedic center SANTY
* Patient with an MRI performed ≥ 3 weeks after ACL tear
* Affiliated patient or beneficiary of a social security scheme
* French-speaking patient who signed an informed consent

Exclusion Criteria:

* Patient with a surgical history on the affected knee
* Patient with a multi-ligament lesion
* Patient already included in another study
* Protected patient: adult under guardianship, curatorship or other protection legal, deprived of liberty by judicial or administrative decision
* Patient hospitalized without consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Manual 3D knee reconstruction from MRI and scanner | 1 day
  Mean IoU (Intersection-Over-Union metric)
Manual 3D knee reconstruction from MRI and scanner | 1 day
  DICE coefficient

SECONDARY OUTCOMES:
Manual and AI 3D knee reconstruction from MRI | 1 day
  Mean IoU (Intersection-Over-Union metric)
Manual and AI 3D knee reconstruction from MRI | 1 day
  DICE coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand SONNERY COTTET, MD, Principal Investigator — GCS RAMSAY SANTE
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No